CLINICAL TRIAL: NCT00205829
Title: Bion for Occipital Nerve Stimulation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR-B-(E)-003
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Headaches
Keywords: Chronic headaches; greater occipital nerve stimulation
MeSH Terms: conditions — Headache Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Active Therapy (Experimental): Occipital nerve stimulation (ONS) therapy delivered to a subject implanted with a bion ONS device
  Interventions: Device: battery-powered bion(R) microstimulator system

INTERVENTIONS:
Device: battery-powered bion(R) microstimulator system — Stimulation on from initial activation and on.

SUMMARY:
This is a prospective, single-centre, cross-over study designed to evaluate the safety and efficacy of using the bion, an implantable medical device, for the treatment of chronic headaches. The clinical study is proposed to determine the anticipated adverse event rate and treatment outcomes at the conclusion of the study. Each trial subject will serve as his/her own control.

ELIGIBILITY:
Inclusion Criteria:

1. Be diagnosed with chronic migraine or primary chronic daily headache
2. Have headaches characterized by pain
3. Be 18 years of age or older;
4. Be willing and able to follow all study-related procedures during course of study;
5. Have exhibited refractoriness to two acute medication regimens and two prophylactic medications from two separate preventive classes.

Exclusion Criteria:

1. Have received a botulinum toxin (botox) injection for treatment of headache within the last 90 days;
2. Have previously undergone destructive ganglionectomy
3. Have had a previous surgery in the intended implant area;
4. Have Arnold-Chiari malformation;
5. Have participated within the last 30 days or plan to participate during this study in another device or drug trial;
6. Be pregnant or planning on becoming pregnant during the study period;
7. Have an implanted electrical device (e.g., pacemaker, spinal cord stimulator) that may interfere with this therapy;
8. Demonstrate significant psychological signs, substance abuse symptoms, or behavioral problems on examination and/or history that, in the investigator's judgment, render them inappropriate for the study;
9. Currently require, or be likely to require, diathermy;
10. Have other medical conditions that the investigator believes would confound the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-06; Primary Completion 2007-08 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Demonstrate acceptable rate of adverse events. | Throughout the Study
The primary efficacy measure is a significant reduction in either headache frequency or severity | 4 months Post-Activation Visit

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Goadsby, MD, Principal Investigator — University College London Hospitals
Locations (1):
- University College London - Institute of Neurology, London, United Kingdom